CLINICAL TRIAL: NCT03375723
Title: Effects of Information and Breathing Technique - for Patients With Respiratory Associated Chest Pain in Acute Pulmonary Embolism. A Randomized, Controlled Multicenter Study.
Brief Title: Effects of Information and Breathing Technique - for Patients With Respiratory Pain in Acute Pulmonary Embolism.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FoU in VGR 235991
Record Dates: First submitted 2017-12-06; First posted 2017-12-18 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Pulmonary Embolism
Keywords: Pain measurement; Pain
MeSH Terms: conditions — Pulmonary Embolism; Pain | interventions — Functional Status

STUDY DESIGN:
Intervention Model Description: A randomized, controlled, intervention study. Evaluation of the addition of information and breathing technique for patients with respiratory associated chest pain in acute pulmonary embolism compared to standard care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Information on anatomy and physiology, and breathing technique (Experimental): Information on anatomy and physiology, and breathing technique
  * Information about anatomy
  * Information about physiology
  * Breathing technique
  Interventions: Other: Information on anatomy and physiology, and breathing technique
- Usual care treatment (Active Comparator): Usual care treatment given to patients with respiratory associated pain in acute PE, which is treatment with analgesics. The information on anatomy and physiology in acute PE is the usual information given by the physician at the ward that the patient is treated.
  Interventions: Other: Usual care treatment

INTERVENTIONS:
Other: Information on anatomy and physiology, and breathing technique — The patients in the treatment group receive information about what acute PE is regarding anatomy and physiology, a review of what causes the respiratory associated pain in acute PE and also a review of the breathing technique to manage their respiratory associated pain. The given information is standardized and the patient also receives written information with both text and pictures. Patients in the treatment group will meet the physiotherapist at day 1, 2 and the patients also has an opportunity to see the physiotherapist or talk to her at the phone if there are any questions concerning the study.
  Arms: Information on anatomy and physiology, and breathing technique
Other: Usual care treatment — Usual care treatment given to patients with respiratory associated pain in acute PE, which is treatment with analgesics. The information on anatomy and physiology in acute PE is the usual information given by the physician at the ward that the patient is treated.
  Arms: Usual care treatment

SUMMARY:
Acute pulmonary embolism (PE) is a serious disease and the third most common cardiovascular disease following myocardial infarction and stroke. The most common symptoms of acute PE are breathlessness and respiratory pain. Although many patients have respiratory pain in acute PE, the treatment of pain is not well described in literature. It is also unclear how long after acute PE the respiratory pain persists. In other conditions with respiratory associated pain, clinical treatment guidelines are available to avoid complications, such as pneumonia, related to impaired respiratory function.

The purpose of this randomized controlled multicenter study is to evaluate the effect of a treatment, in patients with respiratory associated acute PE pain, consisting of information on anatomy and physiology in acute PE and breathing technique in addition to usual care treatment. The above treatment will be compared to conventional treatment in PE with respiratory associated pain, which means treatment with analgesics.

One hundred sixty patients recruited from the Sahlgrenska University Hospital and Alingsås Hospital will participate in the study.

Both groups are examined before and after interventions related to respiratory associated pain, measured with visual analogue scale (VAS), analgesic consumption, lung function measured with Peak Expiratory Flow (PEF), physical disability impairment measured by Disability Rating Index (DRI) and questions about the patients self-efficacy on managing their respiratory associated pain, days hospitalized, pneumonia rate during or after hospitalization, oxygen saturation and patient satisfaction.

Both groups are followed from the inclusion date to 14 days after inclusion through physical visits by the physiotherapist during hospital care and by telephone contact after discharge.

If the positive clinical experience of the information and breathing technique can be confirmed in the study, the method could be spread and used as an easily accessible new treatment method.

DETAILED DESCRIPTION:
Acute pulmonary embolism (PE) is one of the manifestations of venous thromboembolism (VTE) and is a serious and potentially life threatening condition. VTE is the third most common cardiovascular disease after myocardial infarction and stroke, and in the West, with its aging population, a major health problem. In Sweden, the number of diagnosed cases of acute PE is 20-60 per 100,000 inhabitants per year.

The most common symptoms of acute PE are breathlessness and respiratory associated pain. The respiratory pain is an inflammatory pain that originates from the vessels where the embolisms are located. The pain occurs through an irritation of the visceral pleural membrane and creates a sharp, clearly localized pain that increases during deep breathing, coughing and in some cases in motion.

The National Board of Health and Welfare in Sweden´s guidelines for the treatment of venous thromboembolism state that "thrombosis can cause acute pain and the disease may generate anxiety especially in respiratory symptoms". It is unclear how long the pain persists. In a previous study of our research group, 30% of patients had residual respiratory associated pain at discharge after being treated for acute PE.

Although many patients have respiratory associated pain in acute PE, there are no clear description of how this pain should be treated in current guidelines internationally and nationally in Sweden.

Evidence exists that patients with respiratory pain for example after surgery or after costae fracture, should use breathing exercises to increase their ventilation and reduce the risk of complications such as pneumonia and atelectasis.The exercise consists of deep breathing exercise focusing on exhalation with a positive expiratory pressure-device or breathing exercise focused on inhalation with an inhalation spirometer, which has been shown to reduce pleural pressure, increase lung expansion and provide better gas exchange. As far as we know, there are currently no studies on the treatment of respiratory related pain in acute PE.

The aim of the study is to evaluate the effect of a treatment method in addition to the usual care treatment for patients with respiratory associated pain in acute PE. The treatment consists of information and breathing technique and is compared in the usual care treatment for patients with respiratory associated pain, which means treatment with analgesics.

Patients are recruited from wards at the Medical, Cardiovascular and Oncology Clinics at Sahlgrenska University Hospital and Alingsås Hospital. Patients are identified and recruited in the ward they are cared for by physical therapist on duty. All requested patients receive oral and written patient information and shall give their informed consent before inclusion in the study. The patient is randomized via closed-envelope randomization by an independent person to participation in either treatment group or control group.

Intervention Upon inclusion, all patients receive detailed written and oral information about the study and how to register in the study protocols by the physiotherapist at the hospital where they are being treated. The patients randomized to the treatment group also receive information on anatomy and physiology in acute PE as well as the breathing technique.

The information that the patient in the treatment group receives is information about what acute PE is regarding anatomy and physiology, a review of what causes the respiratory associated pain in acute PE and also a review of the breathing technique to manage their respiratory associated pain.

Both groups are informed about using the analgesics they need, but the treatment group is instructed to primarily use breathing techniques to cope with the pain.

A protocol about the information on anatomy and physiology as well as about the breathing technique is used to ensure that the physiotherapists in the study provide the same standardized information to the patients. Written information on anatomy and physiology and breathing technique is also given to patients in the treatment group so that he/she can control that he/she uses the breathing technique correctly when the physiotherapist is not present.

During the time hospitalized, the patient is visited by the physiotherapist day 1, day 2 and at the day for discharge. If the patient has questions or needs support concerning the breathing technique between visits, visits by the physiotherapist or telephone contact are possible. All patients are monitored for 14 days from the inclusion date regarding pain, analgesic consumption and breathing technique training for the patients in the treatment group.

A follow-up with the patient takes place on day 7 and day 15, if the patient is discharged from hospital, this follow-up is done over the phone. On day 15, the patients send the study protocols to the physiotherapist responsible for the study.

Data will be analyzed with Statistic Package for the Social Sciences (SPPS). Both parametric and non-parametric statistics will be used. Data is presented as mean, standard deviation or median and range depending on the variable type. For comparisons between groups in quantitative variables, paired t-tests and ANOVA with post-hoc analyzes will be used. For qualitative variables, Mann Whitney U test and Kruskal-Wallis test will be used. Variables that are dichotomous will be analyzed by Chi2 test or Fisher's exact test.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 80 years of age that understands oral and written instructions in Swedish
* Presence of respiratory associated chest pain from a verified acute pulmonary embolism.
* Presence of respiratory associated pain after moving from a lying to a seated position and taken three deep breaths
* At the time of assessment of pain estimate his/hers pain to >30 mm on the Visual Analogue Scale.

Exclusion Criteria:

* Serious physical illness that includes thorax ie. trauma, lung cancer or rheumatological disease
* Serious non-treated psychiatric disease including psychiatric and psychological disease which are the main cause to the patients pain
* Severe alcohol- or substance abuse
* Treatment with opioids before the diagnosis of acute pulmonary embolism. -Prolonged cancer/ non-cancer related pain.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Respiratory associated pain estimated with Visual Analogue Scale (VAS). | Daily during the whole study period of 14 days.
  Self-assessment of pain intensity of respiratory associated pain according to VAS (scale 0-10, "no pain" vs. "worst possible pain"). Pain intensity is estimated by the patient after moving from lying to sitting and taking three deep breaths. Estimation once a day of average pain during the day is estimated throughout the entire study period. VAS is an instrument for self-estimation of pain which in studies has proven to be both valid and reliable in estimating acute pain.
Analgesic consumption | Daily during the whole study period of 14 days.
  Daily consumption of analgesics is recorded in the study protocol via the patient record. When the patient is discharged from hospital, the patient registers what type of analgesics the patient has taken and in what amount in the study protocol.

SECONDARY OUTCOMES:
Frequency use of breathing technique. | Daily during the whole study period of 14 days.
  Patients in the treatment group register the frequency of the use of the breathing technique during the whole day.
  The registration of breathing techniques is divided into sections where, 1-3 times, 4-6 times, 7-10 times or more than 11 times a day, are the different options. Measurement once a day throughout the study period.
Lung function measurement with Peak Expiratory Flow (PEF) | Measurement takes place on the day of inclusion and at the day for discharge from hospital. If the patient is not discharged within 14 days, the measurement takes place at day 14.
  A measurement of the patient's ability to breathe out his/hers air three times is tested using a PEF-device. The measurement is an objective measure of the patient's ability to create a maximum airflow value during expiration, which may identify possible airway obstruction.
Questions about patients self-efficacy on coping with pain | The questions are asked by a protocol on the day of inclusion, day 7 and day 14.
  Patients will respond to three claims of confidence in their own ability to cope with their pain.
  The claims are rated from "Not sure" to "Absolutely safe" on a 100-millimeter horizontal line and are:
  * How sure are you on your ability to reduce your respiratory associated pain significantly?
  * How sure are you that you can achieve a small to moderate decrease in your respiratory associated pain by means other than increased medication?
  * How sure are you that you can achieve a significant reduction in your respiratory associated pain by means other than increased medication? The questions used are chosen from a scale of self-efficacy and are used exploratively to seek more knowledge of the patients own experience of managing the pain associated with acute LE.
Functional index estimated with Disability Rating Index (DRI). | Estimation takes place on the day of inclusion, day 7 and day 14.
  The patient estimates his/hers perceived physical impairment in performing twelve different physical activities from making simpler activities to exercise physically strenuous activities.
  The patient estimates his ability to perform the activity from "manage without difficulty" to "unable to perform" on a horizontal line that is 100 mm long. DRI is an instrument commonly used for patients with musculoskeletal disabilities. For this patient group, DRI has proven to have both high validity and reliability. DRI has also been used for patients with stable coronary artery disease and has also demonstrated good reliability in the assessment of physical function.

OTHER OUTCOMES:
Number of Days hospitalized | Registration of the outcome takes place at the day for discharge from hospital with a maximal admission time of 14 days.
  Registration on how many days the patient has been admitted to hospital care due to acute pulmonary embolism.
Pneumonia frequency | The patient is asked if he/she have had a pneumonia after falling ill with acute pulmonary embolism. The question is asked at day 14 over the telephone through a Day-14-follow-up-protocol.
  The rate of patients that develops a pneumonia after having acute pulmonary embolism.
Oxygen saturation of the blood | Daily, once a day during hospitalization. If the time hospitalized exceeds 14 days then the last day for registration is day 14.
  Registration of the patients oxygen saturation by a puls oximeter device.

CONTACTS AND LOCATIONS:
Overall Officials: Monika Fagevik Olsén, Professor, Principal Investigator — Göteborg University
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided